CLINICAL TRIAL: NCT01446211
Title: Randomised, Evaluator-Blinded, Multicentre, International, Parallel-Group, Active-Controlled Clinical Trial of Gusperimus Versus Conventional Therapy in Relapse of Granulomatosis With Polyangiitis (Wegener's Granulomatosis) SPARROW Study - SPAnidin in Relapsing GRanulomatosis With POlyangiitis Wegener's Granulomatosis)
Brief Title: Clinical Study Comparing the New Immunosuppressive Drug Gusperimus With the Conventional Treatment in Wegener's Granulomatosis
Acronym: SPARROW
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Change of design consideration
Sponsor: Nordic Pharma SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO005-NK103; 2011-001219-30 (EudraCT Number)
Record Dates: First submitted 2011-09-20; First posted 2011-10-05 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-01

CONDITIONS: Wegeners Granulomatosis
Keywords: gusperimus; Wegeners granulomatosis; relapse
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Recurrence | interventions — gusperimus; Glucocorticoids; Azathioprine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test group - gusperimus (Experimental): Both severity subgroups (severe and non-severe) will be treated with gusperimus + glucocorticoids.
  Interventions: Drug: Gusperimus + glucocorticoids
- Control group (Active Comparator): The severe subgroup will receive a course (13 - 22 weeks) of cyclophosphamide followed by methotrexate + glucocorticoids. Patients intolerant to methotrexate and patients with impaired renal function will receive azathioprine + glucocorticoids.
  The non-severe subgroup will receive methotrexate + glucocorticoids(or azathioprine + glucocorticoids for those previously intolerant to methotrexate or with impaired renal function).
  Interventions: Drug: cyclophosphamide followed by methotrexate (azathioprine) + glucocorticoids or methotrexate (azathioprine) + glucocorticoids

INTERVENTIONS:
Drug: Gusperimus + glucocorticoids — Both severity subgroups will be treated with gusperimus + glucocorticoids up to 12 months.
  Arms: Test group - gusperimus
Drug: cyclophosphamide followed by methotrexate (azathioprine) + glucocorticoids or methotrexate (azathioprine) + glucocorticoids — Severe subgroup: will receive intravenous cyclophosphamide pulses for at least 13 weeks and 22 weeks at maximum, followed by methotrexate + glucocorticoids after achieving a response with BVAS ≤ 2. Patients intolerant to methotrexate and patients with impaired renal function will receive azathioprine + glucocorticoids .
  Non-severe subgroup: will receive methotrexate + glucocorticoids (or azathioprine + glucocorticoids for those previously intolerant to methotrexate or with impaired renal function).
  Arms: Control group

SUMMARY:
The aim of the study is to assess the efficacy (superiority testing) of gusperimus compared to conventional treatment in patients with a relapse of Wegener Granulomatosis with or without ongoing steroids, and/or immunosuppressive therapy. Further, to evaluate the safety and quality of life of gusperimus treatment compared to standard treatment in patients with relapse of Wegener Granulomatosis receiving glucocorticoids.

DETAILED DESCRIPTION:
Wegener Granulomatosis without treatment is life-threatening. The standard treatment with corticosteroids and cyclophosphamide is usually effective at controlling active disease. However, disease relapse is frequent and requires increased exposure to these toxic drugs. In other patients initiation or continuation of these standard drugs is contraindicated due to intolerable side effects. No well-established therapy is available for relapsing patients. They may suffer severe organ damage due to progressive disease, or may die. The proposed indication for gusperimus is the treatment of relapsing Wegener Granulomatosis. The aim of therapy with gusperimus is to induce and maintain remission thereby avoiding further cyclophosphamide and reducing corticosteroid exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of Wegener's Granulomatosis (WG) according to the American College of Rheumatology classification criteria.
2. Diagnosis of WG at least 6 months before entry and initial induction therapy with a combination of Glucocorticoids and an immunosuppressive (Cyclophosphamide or Methotrexate) or rituximab.
3. Relapse of WG with or without ongoing Glucocorticoids, and/or immunosuppressive therapy with Azathioprine/Mycophenolate Mofetil/Methotrexate or Leflunomide. The minimum disease activity is defined by the presence of one new/worse major or three new/worse minor BVAS (version 3) items.
4. Patients between 18 - 75 years.
5. Medically acceptable and reliable contraception method during the study course. (Women should not become pregnant for at least 6 months after Cyclophosphamide treatment).
6. Written informed consent for study participation given by the patient.
7. Patients able and prepared to self-administer the study medication or having a relative/third person able to do it.
8. Ability to read, understand and record information required by protocol

Exclusion Criteria:

1. Other multi-system autoimmune disorders, including systemic lupus erythematosus and anti-Glomerular Basement Membrane disease.
2. Systemic vasculitis due to a viral infection.
3. Cyclophosphamide therapy intolerance, hypersensitivity or contraindication to Cyclophosphamide (active substance or any of the excipients) in patients with severe relapse of WG.
4. Hypersensitivity or contraindication to

   * Spanidin (active substance or any of the excipients) or
   * both Methotrexate (active substance or any of the excipients) and Azathioprine(active substance or any of the excipients) or
   * methylprednisolone, prednisolone or other corticosteroids (active substance or any of the excipients).
5. Underlying medical conditions, which in the opinion of the Investigator place the patient at an unacceptable risk level for participating in a study.
6. Previous randomisation in this study.
7. Cyclophosphamide , intravenous immunoglobulin, anti-cytokine biologic therapies, plasma exchange or Abatacept in the three months prior to entry to the trial. Rituximab, Alemtuzumab or stem cell transplantation is not permitted in the six months prior to entry to the trial.
8. Previous treatment with gusperimus.
9. Participation in another clinical trial with investigational drugs within the last 3 months before screening or during the present trial period.
10. Pregnant or breast-feeding females.
11. Active bacterial/viral infection (Human Immunodeficiency Virus, Hepatitis B, Hepatitis C, Tuberculosis).
12. Patients with Glomerular Filtration Rate (eGFR) < 15 mL/min/1.73m2.
13. Alanine transaminase (ALT), Aspartate aminotransferase (AST), bilirubin, and Alkaline phosphatase (ALP) levels above 2 x the upper normal limit.
14. Inadequate bone-marrow function: White Blood Cells (WBC) < 4000/mm3, haemoglobin < 8 g/dL, neutrophils < 2500/mm3, platelets < 100 000/mm3.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Response rate | 52 weeks
  The primary efficacy variable is the rate of patients showing a response, with the level of disease activity Birmingham Vasculitis Activity Score (BVAS) ≤ 2, within 24 weeks of trial entry, which is maintained without relapse until the end of the trial (Week 52).
  The primary efficacy endpoint includes:
  i) Remission - defined as the complete absence of active clinical disease, i.e. a BVAS score of 0, for at least two months on a stable prednisone dose of ≤ 10 mg/day.
  ii) Low activity Disease State - persistence of up to two minor BVAS items (BVAS ≤ 2).

SECONDARY OUTCOMES:
Time to response | From the date of study entry until the first occasion that BVAS is ≤ 2, assessed up to 52 weeks
  Time to response (response is defined as the time from study entry to the first occasion that BVAS is ≤ 2, and there has been adherence to the steroid reduction protocol)
Response duration | From the date of response with BVAS≤2 until relapse, assessed up to 48 weeks
  Response duration defined as time from response with BVAS≤2 to relapse (relapse is defined as the return or first occurrence of one major and/or three minor BVAS items)
Frequency of severe relapses | Up to 52 weeks
  Frequency of severe relapses (defined as at least one major BVAS item)
Vasculitis Damage Index (VDI) score change | 12 months
  VDI score change from baseline to month 12
Glomerular Filtration Rate (eGFR) change | 12 months
  eGFR change from baseline to month 12 in all patients and in a subgroup defined as having a baseline eGFR ≤ 60mL/min (i.e. renal impairment at baseline)
Frequency of Adverse Events (AEs) and Serious Adverse Event (SAEs) | Up to 52 weeks
  Frequency of AEs and SAEs. (Total number of AEs per group according to AE category) (Percentage of patients in each group with a severe AE)
Frequency of severe infection | Up to 52 weeks
  Frequency of severe infection (a severe infection is defined as an infection that requires intravenous antibiotics or hospitalisation).(Percentage of patients in each group with a severe infection)
Pharmacokinetic parameters at selected sites | 1st day of gusperimus cycles 1, 6 or 7, 12 or 13
  Pharmacokinetic parameters Area Under the plasmaconcentration - time Curve (AUC), Maximum concentration reached in plasma (Cmax), Time to maximum concentration reached in plasma (Tmax) and Elimination half life in plasma (T½) calculated from the measured plasma samples collected at regular time intervals after administration of gusperimus on the first day of three treatment cycles
Short-Form-36 (SF-36) | 6 months
  Pooled physical and mental SF-36 domains change from baseline to month 6
Short-Form-36 (SF-36) | 12 months
  Pooled physical and mental SF-36 domains change from baseline to month 12
Total corticosteroid exposure | Up to 52 weeks
  The total corticosteroid exposure
Questionnaire EQ-5D | 12 months
  Change in EQ-5D between baseline and month 12
Frequency of non-severe relapses | Up to 52 weeks
  Frequency of non-severe relapses (defined as at least 3 minor BVAS items with no major BVAS items).

CONTACTS AND LOCATIONS:
Overall Officials: David Jayne, MD, Principal Investigator — Addenbrookes Hospital, Cambridge, United Kingdom
Locations (1):
- Všeobecná fakultní nemocnice v Praze, Prague, Czechia